CLINICAL TRIAL: NCT06665165
Title: Phase 1, Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Study to Evaluate Safety, Tolerability, PK and PD of Antisense Oligonucleotide AMX0114 Administered to Adult Participants With Amyotrophic Lateral Sclerosis
Brief Title: AMX0114 in Adult Participants With Amyotrophic Lateral Sclerosis
Acronym: LUMINA
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Amylyx Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A114-001
Record Dates: First submitted 2024-10-25; First posted 2024-10-30 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: ALS
Keywords: Amyotrophic Lateral Sclerosis; Sporadic ALS; Motor Neuron Disease; Antisense oligonucleotide; ASO; Calpain-2
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active Treatment: AMX0114 (Experimental): AMX0114 will be administered once every 4 weeks by intrathecal bolus injection for a total of up to 4 doses. Treatment will be administered on Day 1, followed by repeat dosing every 4 weeks at approximately Day 29, Day 57 and Day 85.
  Interventions: Drug: AMX0114
- Placebo (Placebo Comparator): Placebo drug will be administered once every 4 weeks by intrathecal bolus injection for a total of up to 4 doses. Treatment will be administered on Day 1, followed by repeat dosing every 4 weeks at approximately Day 29, Day 57 and Day 85.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: AMX0114 — Antisense oligonucleotides (ASOs) are a type of medicine that treats diseases by intercepting the mRNA messages sent within the cell, resulting in fewer specific proteins being made. AMX0114 is an ASO that targets the mRNA messenger that instructs the body to create a protein called calpain-2. Calpain-2 has been linked to the degeneration and death of neurons in many neurological diseases, including people living with sporadic ALS. AMX0114 is designed to reduce the levels of calpain-2, with the goal of slowing down the process that leads to neuron injury and death.
  Arms: Active Treatment: AMX0114
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a placebo-controlled Phase I study to evaluate the safety, tolerability, pharmacokinetics, and pharmacodynamics of the antisense oligonucleotide (ASO) AMX0114 in adult participants with amyotrophic lateral sclerosis (ALS).

DETAILED DESCRIPTION:
The purpose of this study is to determine how safe and tolerable the investigational drug, AMX0114, is for the treatment of amyotrophic lateral sclerosis (ALS).

AMX0114 is given by intrathecal injection, an injection in the lower back into the spinal canal, also known as lumbar puncture. This clinical trial is designed to test if the treatment is safe and tolerable by monitoring the incidence of adverse events, serious adverse events, dose limiting toxicities (DLTs), and incidence of abnormalities in clinical laboratory assessments, vital signs, physical and neurological examinations, and electrocardiograms (ECGs). This trial will also assess the effects of AMX0114 on biomarkers of ALS, including markers of neuronal death and neuroinflammation.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the purpose and risks of this study, willingness to comply with the study and to provide informed consent in accordance with local laws and regulations.
2. Male or female, at least 18 years of age.
3. Diagnosis of clinically definite or clinically probable ALS, made by a physician who is experienced with management of ALS.
4. Time since onset of first symptom of ALS should be <24 months prior to beginning the study. Date of ALS symptom onset is defined as the onset of weakness (in the limbs, bulbar region, or trunk).
5. If the participant is to be treated with riluzole and/or edaravone before or during the trial, then treatment must be previously started and maintained at a stable regimen for at least 30 days prior to starting the study and through the end of the study.
6. Women of childbearing potential (e.g., not post-menopausal for at least one year or surgically sterile) must agree to use an acceptable birth control method for the duration of the trial and 60 days after the last dose of Study Drug or be of non-childbearing potential.
7. Female participants or female partners of male participants must not be pregnant or plan to become pregnant for the duration of the trial and for up to 90 days after the last dose of Study Drug.
8. Male participants must agree to abstain from sperm donation for the duration of the trial and practice contraception with a female partner, for at least 90 days after last dose of Study Drug.

Exclusion Criteria:

1. Presence of tracheostomy or permanent assisted ventilation.
2. SVC less than 75%.
3. Abnormal liver function defined as aspartate aminotransferase and/or alanine aminotransferase > 3 times the upper limit of normal (ULN) and/or total bilirubin > 1.5 times the ULN (obtained within 4 weeks of first dose) except when a result of Gilbert syndrome.
4. Abnormal renal function defined as estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73m2.
5. Other laboratory abnormalities, including abnormalities in platelet count, international normalized ratio, prothrombin time, and activated partial thromboplastin time.
6. Pregnant women (confirmed by a pregnancy test within 7 days prior to first dose) or women currently breastfeeding.
7. Current or previous clinically significant, unstable medical condition (other than ALS), that in the opinion of the Investigator could affect a participant's safety or ability to comply with the study.
8. Significant abnormalities in physical/neurological examination, vital signs, or electrocardiogram (ECG), which in the opinion of the Investigator could affect the safety of the participant.
9. Presence of unstable psychiatric disease, cognitive impairment, dementia or substance abuse that could affect the participant's ability to provide informed consent or comply with study procedures.
10. Current or previous enrollment in another trial involving use of an investigational therapy, in most cases within 30 days after the last dose of the study drug, prior to starting this study.
11. Current or previous treatment with small interfering ribonucleic acid, stem cell therapy, any ASO or gene therapy.
12. Any contraindications for lumbar puncture or repeated intrathecal injection and/or underlying disorders that could be affected by intrathecal injections.
13. Prior severe reaction or known hypersensitivity to any part of the Study Drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-04-07 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of AMX0114 in adult participants living with ALS | Day 1 - Day 145 (End of Study)
  Incidence of adverse events (AEs), serious adverse events (SAEs) and dose limiting toxicities (DLTs).
  Incidence of abnormalities in clinical laboratory assessments, vital signs, physical and neurological examinations, and electrocardiograms (ECGs).

SECONDARY OUTCOMES:
Evaluate the PK of AMX0114 | Day 1 - Day 145 (End of Study)
  Evaluate PK concentrations, including plasma and CSF levels of AMX0114

OTHER OUTCOMES:
Change from baseline at dosing days and end of study in CSF calpain-2 levels. | Day 1 - Day 145 (End of Study)
Change from baseline at dosing days and end of study in CSF and plasma NfL. | Day 1 - Day 145 (End of Study)
Change from baseline at dosing days and end of study in Amyotrophic Lateral Sclerosis Functional Rating Scale - Revised (ALSFRS - R). | Day 1 - Day 145 (End of Study)
  The ALSFRS-R consists of 12 items across 4 subdomains of function (bulbar, fine motor, gross motor, and breathing) with each item scored on a scale from 0 (total loss of function) to 4 (no loss of function). Total scores range from 0 to 48, with higher scores indicating better function.
Change from baseline at dosing days and end of study in Slow Vital Capacity (SVC). | Day 1 - Day 145 (End of Study)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Amylyx, Study Director — Medical Monitor
Locations (14):
- United States (10):
  - University of California, San Diego, La Jolla, California
  - Georgetown University Hospital Pasquerilla Healthcare Center, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Orlando Regional Medical Center, Orlando Health Neuroscience Institute, Orlando, Florida
  - Massachusetts General Hospital, Healey & AMG Center for ALS, Boston, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Temple University of the Commonwealth System of Higher Education, Philadelphia, Pennsylvania
  - Alliance for Multispecialty Research, LLC, Knoxville, Tennessee
  - Houston Methodist Neurological Institute, Houston, Texas
- Canada (4):
  - University of Calgary, Calgary, Alberta
  - McMaster University, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - McGill University Health Centre - Centre for Innovative Medicine, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Proposals for access to IPD by qualified investigators will be reviewed by an independent review committee. Only the de-identified data elements needed to achieve the specific scientific aims of a proposal as outlined in a pre-specified analysis plan will be provided. Study documents such as protocol, SAP, ICF, and CSR, may be provided, if requested and if needed, to conduct the specified analyses.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: TBD: proposals for access to IPD will be reviewed after data is used in regulatory approval in all major countries or regions where filing is planned or after publication, whichever is latest. Exact timing is not currently known.
Access Criteria: Access to IPD will be granted to qualified investigators whose proposed use of the data has been approved by an independent review committee to achieve the aims in their proposal.